CLINICAL TRIAL: NCT01419912
Title: Comparison of Soy-milk and Cow Milk Consumption on Inflammatory Factors, Cardiovascular Factors ,Renal Factors, Fibrinolytic Indice and Oxidative Stress Among Type-2 Diabetic Patients With Nephropathy Stage 1 and 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Model: Crossover
Other Study IDs: soymilk and nephropathy
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-01

CONDITIONS: Inflammation; Oxidative Stress; Fibrinolytic Markers; Blood Pressure and Cardiorenal Risk Factors
MeSH Terms: conditions — Inflammation | interventions — Soy Milk; Milk

ARMS (2):
- soy milk (Experimental)
  Interventions: Dietary Supplement: soy milk
- cow's milk (Experimental)
  Interventions: Dietary Supplement: cow's milk

INTERVENTIONS:
Dietary Supplement: soy milk
  Arms: soy milk
Dietary Supplement: cow's milk
  Arms: cow's milk

SUMMARY:
Soymilk components such as isoflavones, essential fatty acids, phytoesterols, good fats, inositols might have beneficial effects on controlling complication among diabetic nephropathy patients(DN).Most studies in this regard have been examined the effect of soy consumption on cardiorenal risk factors among patients with DN and there are few data about relationship of soy milk consumption and health effect in patients with DN . Therefore, we evaluated the effects of soy milk compared to cow's milk on blood pressure, inflammation, oxidative stress and fibrinolytic markers and cardiorenal risk factors among these patients. This was a cross-over randomized clinical trial which was conducted in Isfahan among diabetic nephropathy patients. Patients were randomly assigned to consume a diet containing cow's milk or a diet in which only one glass of soy milk was substituted; each one for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* adults with (>18y old) diagnosis of type 2 diabetics nephropathy (diabetics subjects that had proteinuria more than 300 mg/day and had GFR more than 90 mL/min )

Exclusion Criteria:

* exclusion criteria included diabetic nephropathy patients that they were pregnant or lactation women
* changing dosage of oral hypoglycemic agents
* insulin therapy
* lipid-lowering medications
* use of hormone replacement therapy
* alcohol and cigarette consumption;allergy or intolerance to soybeans or milk
* presence of breast malignant and avoid of advisory diet

Ages: 28 Years to 81 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
soy milk

SECONDARY OUTCOMES:
HbA1c
creatinin
total cholesterol
insulin
systolic blood pressure
diastolic blood pressure
Malondialdehyde
fibrinogen
Urine creatinine
urine protein
BUN
TNF-α
IL6
FBS
TG
hs-CRP
d-dimer
HDL
LDL

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran

REFERENCES:
- [Derived] Miraghajani MS, Esmaillzadeh A, Najafabadi MM, Mirlohi M, Azadbakht L. Soy milk consumption, inflammation, coagulation, and oxidative stress among type 2 diabetic patients with nephropathy. Diabetes Care. 2012 Oct;35(10):1981-5. doi: 10.2337/dc12-0250. Epub 2012 Jul 11. PMID 22787172